CLINICAL TRIAL: NCT06156410
Title: A Phase I Trial of Cabozantinib (XL184) in Combination With High-dose Ifosfamide in Adults and Children With Relapsed/Refractory Sarcomas (CaIRS Trial)
Brief Title: Cabozantinib With Ifosfamide in Relapsed/Refractory Sarcomas
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Children's Hospital Colorado (Other); Alex's Lemonade Stand Foundation (Industry); Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-019876
Record Dates: First submitted 2023-11-10; First posted 2023-12-05 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Ewing Sarcoma; Osteosarcoma; Sarcomas
Keywords: relapsed; refractory
MeSH Terms: conditions — Sarcoma, Ewing; Osteosarcoma; Sarcoma; Recurrence | interventions — cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Cabozantinib
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib — Participants will receive cabozantinib in combination with high-dose ifosfamide for 5 cycles. If still on study therapy the participants will continue with cabozantinib monotherapy for up to 12 total cycles.

SUMMARY:
The purpose of this study is to better understand how safe and effective the drug cabozantinib in combination with high-dose ifosfamide is in the treatment of children and adults with relapsed/refractory sarcomas.

DETAILED DESCRIPTION:
In this study, the investigators will test the activity of cabozantinib in combination with high-dose ifosfamide as targeted therapy for relapsed/refractory sarcomas. Cabozantinib has been shown to inhibit multiple tyrosine kinases, including potent inhibition of kinases, MET and VEGFR2. Therefore, the goal of this study is to see if Cabozantinib can be used to inhibit MET and VEGFR2, or other tyrosine kinases to drive tumor responses in patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic diagnosis of any sarcoma, including bone and soft tissue sarcomas. Biopsy from current relapse/progression is highly preferred, though will accept tissue from prior relapse/progression or initial diagnosis with approval from the study Principal Investigator or designee.
2. Disease that has progressed on or relapsed after upfront initial therapy, which must have included traditional chemotherapy.
3. Evaluable or Measurable disease, according to Response Evaluation Criteria in Solid Tumors (RECIST v1.1), within 21 days of enrollment.
4. Age, within the following parameters by cohort:

   1. Phase I dose-finding cohort: age 12 to 40 years at the time of enrollment.
   2. Phase I dose-confirmation cohort: age 5 to < 12 years at the time of enrollment.
5. Body surface area (BSA): > 0.35 m2.
6. Performance status: Lansky play (< 16 years of age) or Karnofsky (> 16 years of age) of ≥ 50, corresponding to Eastern Cooperative Oncology Group (ECOG) categories < 2.
7. Prior toxicity: recovery to baseline or grade < 1, as per the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 (v5.0), from all acute toxicities, unless adverse events (AE) are clinically non-significant (i.e. alopecia) or controlled on supportive care (i.e. nausea/vomiting, hypothyroidism).
8. Able to swallow tablets whole.
9. Hematopoietic function:

   1. Absolute neutrophil count > 1,000/uL (without hematopoietic growth factor within the time frame noted below).
   2. Hemoglobin > 8 g/dL (without transfusion in the last 7 days).
   3. Platelets > 100,000/uL (without transfusion in the last 7 days).
10. Renal function:

    1. Normal renal function determined by one of the following means (even if others are outside of normal range): 1) serum creatinine < 1.5 x upper limit of normal (ULN) for age; 2) cystatin C within normal limits; 3) nuclear medicine glomerular filtration rate (GFR) within normal limits, or 4) calculated creatinine clearance of > 70 mL/min/1.73 m2 (≥ 1.17mL/sec)
    2. Urine protein/creatinine ratio (UPCR) ≤ 1 mg/mg (≤ 113.2 mg/mmol), or 24-hour urine protein ≤ 1 g.
11. Hepatic function:

    1. Total bilirubin < 1.5 x ULN (for subjects with Gilbert's disease < 3.0 x ULN).
    2. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase (ALP) ≤ 3 x ULN (ALP ≤ 5 x ULN is allowed with documented bone metastases). For the purpose of this study, the ULN for ALT is defined as 45 IU/L.
    3. Serum albumin > 2.8 g/dL.
    4. Prothrombin time (PT) and partial thromboplastin time (PTT) < 1.3 x ULN.
12. Sexually active fertile subjects and their partners must agree to use medically accepted methods of contraception (i.e. barrier methods, including male condom, female condom, or diaphragm with spermicidal gel) during the course of the study and for 4 months after the last dose of study treatment.
13. Female subjects of childbearing potential must not be pregnant at screening. Female subjects are considered to be of childbearing potential unless one of the following criteria are met:

    1. Pre-pubertal by tanner staging, defined as Tanner stage 1 or 2.
    2. Documented permanent sterilization (i.e. hysterectomy, bilateral salpingectomy, or bilateral oophorectomy). Documentation of permanent sterilization or postmenopausal status may include review of medical records, medical examinations, or medical history interview by study site.

Exclusion Criteria:

1. Radiographic evidence of tumor invading major blood vessels, or endotracheal or endobronchial tumor.
2. Radiographic evidence of tumor invading the gastrointestinal tract, including esophagus, stomach, small or large bowel, rectum, or anus.
3. Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy or surgery (including radiosurgery) and stable for at least 4 weeks prior to enrollment after radiotherapy or major surgery (i.e. removal or biopsy of brain metastasis). Eligible subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of enrollment.
4. Prior progression/relapse with cabozantinib. Prior therapy with cabozantinib without progression/relapse and prior use of other multi-tyrosine kinase inhibitors is allowed.
5. Prior therapy with high-dose ifosfamide (> 10 g/m2/cycle) at any point.
6. Any small molecule inhibitor therapy within 5 half-lives of the drug or 14 days, whichever is shorter, before enrollment.
7. Myelosuppressive chemotherapy within 14 days before enrollment.
8. Autologous bone marrow transplant (auto-BMT) within 42 days before enrollment.
9. Immunotherapy, including chimeric antigen receptor T-cells (CAR-T), within 21 days before enrollment.
10. Small port radiation therapy within 14 days before enrollment. Substantial bone marrow radiation (i.e. > 50% of the pelvis) or craniospinal radiation within 4 weeks before enrollment. Subjects with any clinically relevant ongoing complications from prior radiation therapy should not be treated with cabozantinib until these complications have resolved.
11. Major surgery (i.e. abdominal surgery; excluding intracranial surgery as noted above) within 14 days before enrollment. Minor surgeries (including mediport or tunneled catheter placement; excluding needle biopsy for tumor sampling or peripherally inserted central catheter placement) within 10 days before enrollment. Subjects must have documented complete wound healing from major surgery or minor surgery before enrollment.
12. Hematopoietic growth factors within 7 days (for short-acting growth factor) or 14 days (for long-acting growth factor) before enrollment.
13. Previously identified allergy or hypersensitivity to components of the study treatment formulations. See Table 10 in Section 9.1.4 for components of cabozantinib.
14. History of clinically significant hemorrhagic cystitis, defined as grade > 3 non-infectious cystitis, associated with antineoplastic agents.
15. Any medications that are strong CYP3A4 inducers or inhibitors or medications definitely known to cause QTc prolongation.
16. Concomitant anticoagulation with coumarin agents (i.e. warfarin), direct thrombin inhibitors (i.e. dabigatran), certain direct factor Xa inhibitors (betrixaban), or platelet inhibitors (i.e. clopidogrel). Allowed anticoagulants are the following:

    1. Prophylactic use of low-dose aspirin for cardio-protection (per local applicable guidelines) and low-dose low molecular weight heparins (LMWH).
    2. Therapeutic doses of LMWH and certain direct factor Xa inhibitors (rivaroxaban, edoxaban, apixaban) in subjects without known brain metastases who are on a stable dose of the anticoagulant for at least 1 week before enrollment without clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor.
17. Cardiovascular disease, including:

    1. Class III or IV congestive heart failure (New York Heart Association grading).
    2. Congenital prolonged QT syndrome, clinically significant cardiac arrhythmia, or prolonged corrected QT (QTc) within 14 days before enrollment.
    3. Uncontrolled hypertension, defined as sustained blood pressure > 95th percentile for age, height, and gender for pediatric subjects and > 140/90 mmHg for adult subjects, despite optimal antihypertensive treatment.
    4. Stroke, transient ischemic attack (TIA), myocardial infarction (MI), unstable angina pectoris, or other ischemic or thromboembolic event (excluding those associated with a central line) within 6 months before enrollment.
18. Gastrointestinal disease, including:

    1. Active peptic ulcer disease, inflammatory bowel disease (Crohn's disease, ulcerative colitis), diverticulitis, cholecystitis, symptomatic cholangitis, appendicitis, or acute pancreatitis.
    2. Acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction.
    3. Intra-abdominal abscess within 6 months before enrollment. Complete healing of an intra-abdominal abscess must be confirmed before enrollment.
    4. Any other condition associated with a high risk of perforation, fistula formation, or potential for decreased absorption of cabozantinib, such as tumors invading the GI tract and ongoing visceral complications from prior radiation therapy.
19. Bleeding conditions, including:

    1. Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (i.e. pulmonary hemorrhage) within 12 weeks before enrollment.
    2. Radiographic evidence of acute intracranial hemorrhage. In the absence of clinical symptoms, a baseline CT/MRI brain need not be obtained.
20. Any other active malignancy at time of enrollment or diagnosis of another malignancy within 3 years prior to enrollment that requires active treatment, except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.
21. Other clinically significant disorders that would preclude safe study participation, including:

    1. Cavitating pulmonary lesion.
    2. Serious non-healing wound/ulcer/bone fracture.
    3. Uncompensated/symptomatic hypothyroidism.
    4. Moderate to severe hepatic impairment (Child-Pugh B or C).
    5. Recipient of solid organ transplant, known human immunodeficiency virus (HIV) seropositivity, and other non-treatment related immunodeficiencies.
    6. Severe or uncontrolled infection or systemic disease.
    7. Inadequate electrolyte balance, defined as abnormal levels of serum potassium, calcium, magnesium, and phosphorous and causing clinically significant symptoms, acid-base disturbances, or changes in ECG.
22. Women who are currently pregnant or breastfeeding.

Ages: 5 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose/recommended phase II dose (MTD/RP2D) of cabozantinib | Upon completion of accrual to phase 1 cohort, approximately 1 year
  Toxicity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 (v5.0).

SECONDARY OUTCOMES:
Toxicity profile | Upon completion of trial, approximately 1 year
  Define and describe the toxicity profile (grade 2 and above) of cabozantinib administered in combination with high-dose ifosfamide using Common Terminology Criteria for Adverse Events (CTCAE).
Dose-limiting toxicities (DLT) | After two cycles of treatment, average 56 days (one cycle is 28 days)
  Define and describe the dose-limiting toxicities (DLT) of cabozantinib administered in combination with high-dose ifosfamide using Common Terminology Criteria for Adverse Events (CTCAE).
Antitumor activity Ewing sarcoma | 6 months
  Evaluate the antitumor activity of cabozantinib administered in combination with high-dose ifosfamide for relapsed/refractory Ewing sarcoma using the Response Criteria for Patients with Solid Tumors (RECIST) scale. Disease progression will be measured periodically while on study.
Antitumor activity osteosarcoma | 6 months
  Evaluate the antitumor activity of cabozantinib administered in combination with high-dose ifosfamide for relapsed/refractory osteosarcoma using the Response Criteria for Patients with Solid Tumors (RECIST) scale. Disease progression will be measured periodically while on study.
Antitumor Activity Relapsed/Refractory Sarcomas | 6 months
  Evaluate the antitumor activity of cabozantinib administered in combination with high-dose ifosfamide for relapsed/refractory sarcomas using the Response Criteria for Patients with Solid Tumors (RECIST) scale. Disease progression will be measured periodically while on study.

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Laetsch, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (4):
- United States (4):
  - University of California San Francisco, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Children's Hospital of Philadelphia, as the sponsor and lead site for this trial, will have access to all participant data throughout the study.
  Certain biological samples will be sent to the University of Colorado for processing and analysis.
Supporting Information: Study Protocol, ICF
Time Frame: Participant data will be sent between sites as required by protocol. Sites will all share data with Children's Hospital of Philadelphia and University of Colorado. Data can be accessed and used by the sites for the duration of the study and data analysis period.
Access Criteria: Must be a Children's Hospital of Philadelphia (CHOP) Institutional Review Board (IRB) approved site of the study.